CLINICAL TRIAL: NCT06185972
Title: Novel Magnetic Resonance Imaging-Guided Ultrasound-Stimulated Microbubble Radiation Treatment for Patients With Chest-Wall and Locally Advanced Breast Cancer-Phase II
Brief Title: Novel Magnetic Resonance Imaging-Guided Ultrasound-Stimulated Microbubble Radiation Treatment for Patients With Chest-Wall and Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Terry Fox Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5768
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Focused Ultrasound; Breast Cancer; Microbubbles
MeSH Terms: conditions — Breast Neoplasms | interventions — perflutren; Microbubbles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Treatment Arm (Experimental): All biopsy confirmed breast cancer patients undergoing MRI-guided ultrasound-stimulated microbubble treatment plus radiation therapy
  Interventions: Drug: Definity; Device: Sonalleve Focused Ultrasound Device

INTERVENTIONS:
Drug: Definity — Stimulation of Definity microbubbles using Sonalleve device within tumour vasculature
  Other Names: Microbubbles
Device: Sonalleve Focused Ultrasound Device — Sonalleve Focused Ultrasound Device

SUMMARY:
The objective of this study is to demonstrate the efficacy and response of novel Magnetic Resonance Imaging (MRI)-guided ultrasound stimulated microbubble treatment to enhance radiation effects in humans receiving external beam radiotherapy delivered using a LINAC (linear accelerator) radiation therapy device.

DETAILED DESCRIPTION:
The approach uses relatively low-power ultrasound, operating with lower power levels than high intensity focused ultrasound and ultrasound-based hyperthermia techniques, delivered on the Sonalleve platform. The tumour will be sonicated before the radiation to enhance the effect of therapy. The technique is spatially targeted and stimulates microbubbles using low-power ultrasonic fields in the tumour location only. The primary aim is to evaluate tumour response to MRg-FUS + MB and radiation, as measured radiologically or clinically within the treated therapeutic target regions.The secondary aim of this research is to evaluate early and late effect profiles of MRI- guided ultrasound stimulated microbubble treatment and radiation in patients with inoperable breast/chest wall tumours or LABC at 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 1 year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* All biopsy-confirmed invasive ductal, invasive lobular and other rare histologic types of carcinoma.
* Patients with early stage Breast cancer, or LABC ; i.e., Stage IIA - IIIC cancers (T2 N0 M0 to Any T, N3, M0) or Stage IV (Any T, Any N, M1) per AJCC guidelines (8th Edition).
* Assessed as indicated, by a multidisciplinary team of treating medical, surgical and radiation oncologist and found suitable for radiation treatment.
* Patient referred for standard palliative radiotherapy or curative radiotherapy, which may include (but are not limited to) any of the following dose regimens: 1) 5-8 Gy in one fraction, 2) 20 Gy in 5 fractions, 3) 30 Gy in 5 fractions, 4) 35 Gy in 5 fractions, 5) 30 Gy in 10 fractions, 6) 40 Gy in 10 fractions, 5) 50 Gy in 20 fractions, 6) 60 Gy in 30 fractions and 7) 66 Gy in 33 fractions, or radiobiologically similar doses.
* Able to understand and give informed consent.
* Weight < 140 kg.
* Target lesion accessible for MRg-FUS+MB procedure.
* Able to communicate sensation during the procedure.
* Creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional upper limit of normal.

Exclusion Criteria:

* Pregnant or lactating women may not participate due to the embryotoxic effects of protocol treatment.
* Unable to have a contrast-enhanced MRI scan - standard of care criteria.
* Patients having received anthracycline or taxane based chemotherapy within the past 5 days.
* Patients intended for surgical management of the target tumour.
* Patients with metallic or breast implants.
* Subjects with connective tissue disorder, musculoskeletal deformity.
* Target lesion causing deep ulceration, bleeding or discharge of the overlying skin.
* A fibrotic scar along the proposed FUS beam path.
* Severe cardiovascular, neurological, renal or hematological chronic disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥ 3.
* Any condition that in the investigator's opinion precludes participation.
* Unable to tolerate required stationary position during treatment.
* Allergy to Definity microbubbles.
* Cardiac disease or unstable hemodynamics including myocardial infarction within six months, unstable angina, congestive heart failure, cardiac shunts, cardiac arrhythmia and cardiac pacemaker.
* Contraindication to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation like cisapride, erythromycin, tricyclic antidepressants, Class IA and III antiarrhythmic agents and some antipsychotics like haloperidol, droperidol, quetiapine, thioridazine, ziprasidone.
* Known QT prolongation = (QTc > 450ms for men or >470ms for women) with cardiac impairment if ECG is requested as per SOC.
* History of bleeding disorder, coagulopathy.
* Severely impaired renal function with estimated glomerular filtration rate < 30ml/min/1.73m2 and/or on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcomes/Endpoint | 3 months
  The primary endpoint is complete response (RECIST 1.1 Criteria) in chest-wall tumours and LABC following MRg-FUS + MB + radiation after a 3 month follow up. Patients will be followed clinically thereafter as part of standard of care.

SECONDARY OUTCOMES:
Secondary Outcomes/Endpoint(s) | 1 year
  The secondary endpoint will be late effect-reported outcomes (at 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 1 year after treatment. A toxicity questionnaire will be used as an outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gregory Czarnota, MD, Ph.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No